CLINICAL TRIAL: NCT06616064
Title: Evaluation of a Procedure for Identification and Brief Intervention of Lifestyle Advice Assisted by Application in a Care Setting
Acronym: CliniCAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC23_9738_CliniCAP; 2024-A01631-46 (Other: N°ID-RCB)
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Chronic Disease
Keywords: brief intervention of lifestyle advice
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: personalised feedback and brief motivational; Other: routine lifestyle advice; Other: questionnaire CliniCAP
- Control (Other)
  Interventions: Other: routine lifestyle advice; Other: questionnaire CliniCAP

INTERVENTIONS:
Behavioral: personalised feedback and brief motivational — personalised feedback and brief motivational
  Arms: Experimental
Other: routine lifestyle advice — routine lifestyle advice
Other: questionnaire CliniCAP — questionnaire CliniCAP

SUMMARY:
Chronic diseases share similar risk factors associated with four daily behaviours: unbalanced diet, sedentary lifestyle (physical inactivity and time spent sitting down), smoking and alcohol consumption. These diseases are responsible for 74% of deaths worldwide. Despite the frequency with which practitioners witness these bad habits in their patients, little time is devoted to lifestyle advice during medical visits, and even less to using effective techniques to discuss their behaviour. Yet medical and paramedical consultations could be an essential educational opportunity to promote a healthy lifestyle. But advice is often limited during medical check-ups, due to a lack of time and suitable tools, and is often focused on a particular risk factor. To date, there is no procedure for screening and behavioural intervention to deal with harmful lifestyle habits in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Treated for a stabilised chronic disease OR person treated for localised cancer, after the end of heavy treatment during the follow-up period within 5 years of the date of diagnosis of the cancer.
3. Contactable by telephone
4. Affiliated to a social security scheme
5. Having signed a free, informed and written consent.

Exclusion Criteria:

1. Requiring psychiatric assessment
2. Suffering from eating disorders
3. Undergoing dietetic treatment or therapeutic education for dietetic purposes (at least two consultations at the same facility in the previous year)
4. Suffering from a life-threatening condition within 5 years
5. Suffering from a disabling condition (reduced activity with major restrictions)
6. Unable to read
7. Taking part in another psycho-behavioural nutritional intervention study
8. Protected person (adult subject to legal protection (safeguard of justice, curatorship, guardianship), person deprived of liberty, pregnant woman (declaratory), breast-feeding woman and minor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of green criteria on application feedback | between Day 0 and Month 1
  The green criterioa corresponds to good compliance with health recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Romain Moirand, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France